CLINICAL TRIAL: NCT01822522
Title: Phase I Trial of Cabozantinib (XL184) for Advanced Solid Tumors in Persons With HIV Infection
Brief Title: Cabozantinib S-Malate in Treating Patients With Advanced Solid Tumors and Human Immunodeficiency Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00740; NCI-2013-00740 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-087; AMC-087 (Other: AIDS Malignancy Consortium); AMC-087 (Other: CTEP); U01CA121947 (NIH); UM1CA121947 (NIH)
Record Dates: First submitted 2013-04-01; First posted 2013-04-02 (Estimated); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Advanced Malignant Solid Neoplasm; HIV Infection; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm; Unresectable Solid Neoplasm
MeSH Terms: conditions — HIV Infections; Neoplasm Metastasis | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: In this study, cabozantinib doses were escalated within 3 strata defined by the participant's antiretroviral regimen
Oversight: Data Monitoring Committee: No

ARMS (6):
- Stratum A Treatment (cabozantinib s-malate): 20 mg/day (Experimental): Patients receive cabozantinib s-malate 20 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  This arm includes patients who are on ritonavir-boosted or cobicistat-boosted antiretroviral regimens
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Stratum A Treatment (cabozantinib s-malate): 40 mg/day (Experimental): Patients receive cabozantinib s-malate 40 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  This arm includes patients who are on ritonavir-boosted or cobicistat-boosted antiretroviral regimens
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Stratum A Treatment (cabozantinib s-malate): 60 mg/day (Experimental): Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  This arm includes patients who are on ritonavir-boosted or cobicistat-boosted antiretroviral regimens
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Stratum B Treatment (cabozantinib s-malate): 60 mg/day (Experimental): Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  This arm includes patients who are on efavirenz or etravirine-based antiretroviral regimens
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Stratum B Treatment (cabozantinib s-malate): 100 mg/day (Experimental): Patients receive cabozantinib s-malate 100 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  This arm includes patients who are on efavirenz or etravirine-based antiretroviral regimens
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Stratum C Treatment (cabozantinib s-malate): 60 mg/day (Experimental): Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  This arm includes patients who are on antiretroviral regimens that do not include the agents specified on stratum A or B, or who are not on antiretroviral therapy
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL-184; XL184
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of cabozantinib s-malate in treating patients with solid tumors that have spread to other places in the body and usually cannot be cured or controlled with treatment and human immunodeficiency virus. Cabozantinib s-malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of cabozantinib (XL184) (cabozantinib s-malate) as a single agent in solid tumor participants with human immunodeficiency virus (HIV) infection and to determine the maximal tolerated dose (MTD) in this patient population.

SECONDARY OBJECTIVES:

I. To investigate possible pharmacokinetic interactions between cabozantinib and antiretroviral therapy in persons with HIV infection.

II. To investigate the effects of therapy on participant immune status and HIV viral load.

III. To preliminarily assess objective response rates associated with treatment for commonly represented tumors.

OUTLINE: This is a dose-escalation study.

Patients receive cabozantinib s-malate orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have known HIV infection and histologically confirmed solid malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; any number of prior cancer therapies will be permitted; at least 4 weeks must have elapsed since prior chemotherapy or biological therapy, 6 weeks if the regimen included carmustine (BCNU) or mitomycin C; prior radiation therapy to the thoracic cavity, abdomen, or pelvis must be completed at least 3 months prior to registration; radiotherapy to any other site (including bone or brain metastases) must be completed at least 28 days prior to registration
* Serologic documentation of HIV infection at any time prior to study entry, as evidenced by positive enzyme-linked immunosorbent assay (ELISA), positive western blot, or any other federally approved licensed HIV test; alternatively, this documentation may include a record that another physician has documented that the participant has HIV infection based on prior ELISA and western blot, or other approved diagnostic tests
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL (within 1 week of study entry)
* Absolute neutrophil count >= 1,500/mcL (within 1 week of study entry)
* Platelets >= 100,000/mcL (within 1 week of study entry)
* Total bilirubin=< 1.5 x upper limit of normal (ULN) (within 1 week of study entry) (if, however, the participant has Gilbert's disease or unconjugated hyperbilirubinemia that is considered to be secondary to with atazanavir or indinavir therapy, then the total bilirubin must be =< 3 x ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional upper limit of normal (within 1 week of study entry)
* Creatinine =< 1.5 x ULN (within 1 week of study entry)
* Creatinine clearance >= 50 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal (within 1 week of study entry)
* Hemoglobin >= 9 g/dL (within 1 week of study entry)
* Serum albumin >= 2.8 g/dL (within 1 week of study entry)
* Lipase < 2.0 x ULN and no radiologic or clinical evidence of pancreatitis (within 1 week of study entry)
* Urine protein/creatinine ratio (UPCR) =< 1 (within 1 week of study entry)
* Serum phosphorus >= lower limit of normal (LLN) (within 1 week of study entry)
* Calcium >= LLN (within 1 week of study entry)
* Magnesium >= LLN (within 1 week of study entry)
* Potassium >= LLN (within 1 week of study entry)
* A cluster of differentiation (CD)4+ lymphocyte count > 50/mcL will be required within 2 weeks of study participation
* Women of childbearing potential must have a negative pregnancy test within 7 days before enrollment; women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal; postmenopause is defined as amenorrhea >= 12 consecutive months; note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason
* The effects of cabozantinib on the developing human fetus are unknown; for this reason and because tyrosine kinase inhibitors agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of cabozantinib administration; sexually active participants (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 6 months after the last dose of study drug(s), even if oral contraceptives are also used; all participants of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 6 months after the last dose of study drug
* Participating participants MUST receive appropriate care and treatment for HIV infection, including antiretroviral medications, when clinically indicated and should be under the care of a physician experienced in HIV management; participants will be eligible regardless of antiretroviral medication (including no antiretroviral medication) provided there is no intention to initiate therapy or the regimen has been stable for at least 4 weeks with no intention to change the regimen within 8 weeks following study entry; as study-specific (antiretroviral-based) strata fill, however, only participants who are receiving the therapies eligible for the remaining open strata will be accrued
* Ability to understand and the willingness to sign a written informed consent document
* Participants must in the opinion of the investigator be capable of complying with this protocol

Exclusion Criteria:

* Prior treatment with cabozantinib (XL184)
* The participant has received radionuclide treatment within 6 weeks of the first dose of study treatment
* The participant has received prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within 4 weeks or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment; note: participants with prostate cancer currently receiving luteinizing hormone-releasing hormone (LHRH) or gonadotropin-releasing hormone (GnRH) agonists may be maintained on these agents
* The participant has received any other type of investigational agent within 28 days before the first dose of study treatment
* The participant has not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant adverse events (AEs)
* The participant has a primary brain tumor
* The participant has active brain metastases or epidural disease; participants with brain metastases previously treated with whole brain radiation or radiosurgery or participants with epidural disease previously treated with radiation or surgery who are asymptomatic and do not require steroid treatment for at least 4 weeks before starting study treatment are eligible; participants with treated brain metastasis should not take enzyme-inducing anticonvulsive therapies (EIACDs) within 2 weeks of registration, though non-enzyme inducing anticonvulsive drugs such as levetiracetam are allowed; neurosurgical resection of brain metastases or brain biopsy is permitted if completed at least 3 months before starting study treatment; baseline brain imaging with contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI) scans for participants with known brain metastases is required to confirm eligibility
* The participant has prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test >= 1.3 x the laboratory ULN within 7 days before the first dose of study treatment
* The participant requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or factor xabans (Xa) inhibitors, or antiplatelet agents (e.g., clopidogrel); low dose aspirin (=< 81 mg/day), low-dose warfarin (=< 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted
* The participant requires chronic concomitant treatment with the following strong cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inducers OTHER than antiretroviral agents: dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, primidone, modafinil, and other enzyme inducing anti-convulsant drugs (EIACD), and St. John's wort; use of efavirenz or etravirine is permitted for participants considered for the CYP3A4-inducer based antiretroviral therapy (ART) regimen arm (Stratum B) of the trial; because the lists of CYP3A4 inducers are constantly changing, it is important to regularly consult a frequently-updated list; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product
* The participant requires concomitant treatment with the following inhibitors of CYP3A4:

  * Antibiotics: clarithromycin, erythromycin, telithromycin, troleandomycin
  * Antifungals: itraconazole, ketoconazole, voriconazole, fluconazole, posaconazole
  * Antidepressants: nefazodone
  * Antidiuretic: conivaptan
  * Gastrointestinal (GI): cimetidine, aprepitant
  * Hepatitis C: boceprevir, telaprevir
  * Miscellaneous: Seville oranges, grapefruit, or grapefruit juice and/or pummelos, star fruit, exotic citrus fruits, or grapefruit hybrids); use of any of anti-retrovirals (delavirdine) or protease inhibitors (ritonavir, indinavir, lopinavir/ritonavir, saquinavir, nelfinavir) is permitted; specifically, ritonavir and cobicistat is permitted for participants considered for the CYP3A4-inhibitor based ART regimen arm (Stratum A) of the trial; because the lists of CYP3A4 inhibitors are constantly changing, it is important to regularly consult a frequently-updated list; medical reference texts such as the physicians' desk reference may also provide this information; as part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product
* The participant has experienced any of the following:

  * Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment
  * Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment
  * Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* The participant has radiographic evidence of cavitating pulmonary lesion(s)
* The participant has tumor invading or encasing any major blood vessels
* The participant has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including:

    * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mmHg systolic, or > 90 mmHg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
    * Any history of congenital long QT syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * Unstable angina pectoris
      * Clinically-significant cardiac arrhythmias
      * Stroke (including transient ischemic attack [TIA], or other ischemic event)
      * Myocardial infarction
      * Thromboembolic event requiring therapeutic anticoagulation (note: participants with a venous filter [e.g. vena cava filter] are not eligible for this study)
  * Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

    * Any of the following within 28 days before the first dose of study treatment

      * Active peptic ulcer disease
      * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
      * Malabsorption syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * Abdominal fistula
      * Gastrointestinal perforation
      * Bowel obstruction or gastric outlet obstruction
      * Intra-abdominal abscess; note: complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months before the first dose of study treatment
* Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months before the first dose of study therapy
* Other clinically significant disorders such as:

  * Active infection requiring systemic treatment within 28 days before the first dose of study treatment; participants with HIV infection will be eligible provided they meet the criteria; participants with known hepatitis B infection should be screened for active disease prior to study participation; participants with known hepatitis C infection must not be actively receiving treatment for the infection
  * Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
  * History of organ transplant
  * Concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment
  * History of major surgery as follows:

    * Major surgery within 3 months of the first dose of cabozantinib if there were no wound healing complications or within 6 months of the first dose of cabozantinib if there were wound complications
    * Minor surgery within 1 month of the first dose of cabozantinib if there were no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications
  * In addition, complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of cabozantinib irrespective of the time from surgery
* The participant is unable to swallow tablets that are whole (do not crush or chew or administer via nasogastric [NG]-tube)
* The participant has a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before randomization; note: if initial QTcF is found to be > 500 ms, two additional electrocardiogram (ECGs) separated by at least 3 minutes should be performed; if the a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-06-21 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Missak Haigentz, Principal Investigator — AIDS Malignancy Consortium
Locations (20):
- United States (20):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Center for Clinical AIDS Research and Education, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Louisiana State University, Lafayette, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Street Clinic, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum A - 20 mg/Day: Patients taking either ritonavir-boosted or cobicistat-boosted antiretroviral regimens
  Patients receive cabozantinib s-malate 20 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
- Stratum A - 40 mg/Day: Patients taking either ritonavir-boosted or cobicistat-boosted antiretroviral regimens
  Patients receive cabozantinib s-malate 40 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
- Stratum A - 60 mg/Day: Patients taking either ritonavir-boosted or cobicistat-boosted antiretroviral regimens
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
- Stratum B - 60 mg/Day: Patients taking either efavirenz or etravirine-based antiretroviral regimens
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum B - 100 mg/Day: Patients taking either efavirenz or etravirine-based antiretroviral regimens
  Patients receive cabozantinib s-malate 100 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum C - 60 mg/Day: Patients who are on antiretroviral therapy that does not include agents in stratum A or B, or who were not on antiretroviral therapy
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
Period: Overall Study
Arm/Group | Stratum A - 20 mg/Day | Stratum A - 40 mg/Day | Stratum A - 60 mg/Day | Stratum B - 60 mg/Day | Stratum B - 100 mg/Day | Stratum C - 60 mg/Day
Started | 6 | 7 | 7 | 6 | 3 | 7
Completed | 2 | 6 | 3 | 4 | 3 | 3
Not Completed | 4 | 1 | 4 | 2 | 0 | 4
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0 | 1
Not completed — Death | 3 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Patients who enrolled on the study and whose antiretroviral regimen met the requirements for the appropriate stratum
Groups:
- Stratum A - 20 mg/Day: Patients receive cabozantinib s-malate 20 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Patients in this stratum receive ritonavir-boosted or cobicistat-boosted antiretroviral therapy
- Stratum A - 40 mg/Day: Patients receive cabozantinib s-malate 40 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Patients in this stratum receive ritonavir-boosted or cobicistat-boosted antiretroviral therapy
- Stratum A - 60 mg/Day: Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Patients in this stratum receive ritonavir-boosted or cobicistat-boosted antiretroviral therapy
- Stratum B - 60 mg/Day: Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Patients in this strata receive efavirenz or etravirine-based antiretroviral regimens
- Stratum B - 100 mg/Day: Patients receive cabozantinib s-malate 100 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Patients in this strata receive efavirenz or etravirine-based antiretroviral regimens
- Stratum C - 60 mg/Day: Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Patients in this arm receive antiretroviral therapy that does not include the agents in stratum A or B, or are not on antiretroviral therapy
- Total: Total of all reporting groups
Arm/Group | Stratum A - 20 mg/Day | Stratum A - 40 mg/Day | Stratum A - 60 mg/Day | Stratum B - 60 mg/Day | Stratum B - 100 mg/Day | Stratum C - 60 mg/Day | Total
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 3 | 7 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (14.9) | 48.9 (10.4) | 45.9 (13.0) | 50.5 (6.7) | 48.0 (7.8) | 49.9 (9.2) | 49.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Male | 6 | 6 | 6 | 5 | 3 | 7 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 2 | 1 | 0 | 7
  Not Hispanic or Latino | 4 | 6 | 6 | 4 | 2 | 7 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 4 | 1 | 1 | 4 | 13
  White | 4 | 5 | 2 | 4 | 2 | 3 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 7 | 6 | 3 | 7 | 36

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Will be reported using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The number of participant who experienced an adverse event
Time Frame: Up to 30 days after completion of study treatment. Study treatment was between 1 and 82 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Stratum A - 20 mg/Day: Patients who were on ritonavir-boosted or cobicistat-boosted antiretroviral regiments.
  Patients receive cabozantinib s-malate 20 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
- Stratum A - 40 mg/Day: Patients who were on ritonavir-boosted or cobicistat-boosted antiretroviral regiments.
  Patients receive cabozantinib s-malate 40 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
- Stratum A - 60 mg/Day: Patients who were on ritonavir-boosted or cobicistat-boosted antiretroviral regiments.
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
- Stratum B - 60 mg/Day: Patients who are on efavirenz or etravirine-based antiretroviral regimens.
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
- Stratum B - 100 mg/Day: Patients who are on efavirenz or etravirine-based antiretroviral regimens.
  Patients receive cabozantinib s-malate 100 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
- Stratum C: Patients who are not on the antiretroviral regimens specified in stratum A or B, or who were not on an antiretroviral regimen
  Patients receive cabozantinib s-malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
Arm/Group | Stratum A - 20 mg/Day | Stratum A - 40 mg/Day | Stratum A - 60 mg/Day | Stratum B - 60 mg/Day | Stratum B - 100 mg/Day | Stratum C
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 3 | 7
Participants | 6 | 7 | 7 | 6 | 3 | 7

2. Primary Outcome: Maximal Tolerated Dose (MTD) of Cabozantinib-s-malate
Description: Will be graded according to the NCI CTCAE version 5.0. Dose-limiting toxicity (DLT) will be defined as any cabozantinib s-malate related grade 3 or 4 non-hematologic toxicity including grade 3 nausea and/or vomiting and grade 3 diarrhea despite prophylaxis and/or treatment or any of the following grade 4 hematologic toxicities: thrombocytopenia and neutropenia of any duration (with or without fever or documented infection); additionally, treatment delay of greater than 7 days due to unresolved toxicity or any dose reduction required due to a cabozantinib-related adverse event will be considered a DLT.
Time Frame: Up to 28 days after treatment initiation
Measure: Number; unit: mg/day
Groups:
- Stratum A: Patients who are receiving ritonavir-boosted or cobicistat-boosted antiretroviral therapy.
  Patients receive cabozantinib s-malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
- Stratum B: Patients who are on efavirenz or etravirine-based antiretroviral regimens.
  Patients receive cabozantinib s-malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
- Stratum C: Patients who are on antiretroviral therapy regimens that do not include the agents in stratum A or stratum B, or are not on antiretroviral therapy.
  Patients receive cabozantinib s-malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 20 | 9 | 7
mg/day | 20 | 60 | 60

3. Secondary Outcome: Response Rates
Description: Will be using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors guideline (version 1.1). Binomial proportions and their 95% confidence intervals will be used. Responses are categorized as complete or partial.
Time Frame: Up to 30 days after completion of study treatment. Study treatment was between 1 and 82 weeks. The median number 28-day cycles was 3.5.
Measure: Count of Participants; unit: Participants
Groups:
- Stratum A 20 mg/Day: Patients who were on ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 20 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum A - 40 mg/Day: Patients who were on ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 40 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum A - 60 mg/Day: Patients who were on ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum B - 60 mg/Day: Patients who are on efavirenz or etravirine-based antiretroviral therapy
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum B - 100 mg/Day: Patients who are on efavirenz or etravirine-based antiretroviral therapy
  Patients receive cabozantinib s-malate 100 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum C - 60 mg/Day: Patients who are not on an antiretroviral therapy that includes the agents in stratum A or B, or are not on an antiretroviral therapy.
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
Arm/Group | Stratum A 20 mg/Day | Stratum A - 40 mg/Day | Stratum A - 60 mg/Day | Stratum B - 60 mg/Day | Stratum B - 100 mg/Day | Stratum C - 60 mg/Day
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 3 | 7
Participants | 0 | 0 | 1 | 2 | 0 | 2

4. Secondary Outcome: Human Immunodeficiency Virus (HIV) Viral Load
Description: Detectable HIV viral load at visit 04 (day 22)
Time Frame: Day 22 of treatment
Population: Participants who had HIV viral load measurements at visit 04
Measure: Count of Participants; unit: Participants
Groups:
- Stratum A - 20 mg/Day: Patients that are on ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 20 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum - 40 mg/Day: Patients that are on ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 40 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum A - 60 mg/Day: Patients that are on ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum B - 60 mg/Day: Patients who are on efavirenz or etravirine-based antiretroviral treatment
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum B - 100 mg/Day: Patients who are on efavirenz or etravirine-based antiretroviral treatment
  Patients receive cabozantinib s-malate 100 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum C - 60 mg/Day: Patients who are on an antiretroviral regimen that does not include the agents in stratum A or B, or are not on antiretroviral therapy
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
Arm/Group | Stratum A - 20 mg/Day | Stratum - 40 mg/Day | Stratum A - 60 mg/Day | Stratum B - 60 mg/Day | Stratum B - 100 mg/Day | Stratum C - 60 mg/Day
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 3 | 7
Participants | 3 | 4 | 2 | 3 | 1 | 4

5. Secondary Outcome: CD4+ Cell Counts
Description: Change in CD4 counts from baseline to visit 04
Time Frame: Day 22 of treatment
Measure: Mean (Standard Deviation); unit: cells/mm^3
Groups:
- Stratum A-20 mg/Day: Patients who are ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 20 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum A - 40 mg/Day: Patients who are ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 40 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum A - 60 mg/Day: Patients who are ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum B - 60 mg/Day: Patients on efavirenz or etravirine-based antiretroviral therapy
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum B - 100 mg/Day: Patients on efavirenz or etravirine-based antiretroviral therapy
  Patients receive cabozantinib s-malate 100 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum C - 60 mg/Day: Patients who are on antiretroviral therapy that does not include agents in stratum A or B, or who are not on antiretroviral therapy
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
Arm/Group | Stratum A-20 mg/Day | Stratum A - 40 mg/Day | Stratum A - 60 mg/Day | Stratum B - 60 mg/Day | Stratum B - 100 mg/Day | Stratum C - 60 mg/Day
Number analyzed (Participants) | 3 | 4 | 2 | 3 | 1 | 4
cells/mm^3 | 41.0 (31.2) | 30.0 (45.2) | 64.5 (92.6) | 23.0 (127.6) | 33.0 (0) | -87.5 (17.7)

6. Secondary Outcome: CD8+ Cell Counts
Description: Change in CD8 cell counts from baseline to visit 04.
Time Frame: Day 22 of treatment
Population: Participants with baseline and visit 4 CD8 counts. Absolute CD8 counts were not collected on the study.
Groups:
- Stratum A: Patients who are on ritonvir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum B: Patients who are efavirenz or etravirine-based antiretroviral therapy
  Patients receive cabozantinib s-malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum C: zPatients who are on an antiretroviral regimen that does not include agents in stratum A or B, or who are not on antiretroviral therapy
  Patients receive cabozantinib s-malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Pharmacokinetic Parameters
Description: Cmax at the maximum tolerated dose: 20 mg for stratum A, 60 mg for stratums B and C
Time Frame: Day 1
Population: Participants in stratum with Cmax levels at the maximum tolerated dose: 20 mg for stratum A, 60 mg for stratums B and C
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Groups:
- Stratum A - 20 mg/Day: Patients on ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 20 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum C - 60 mg/Day: Patients on antiretroviral therapy that does not contain the agents in stratum A or B, or who were not on antiretroviral therapy
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
Arm/Group | Stratum A - 20 mg/Day | Stratum B - 60 mg/Day | Stratum C - 60 mg/Day
Number analyzed (Participants) | 5 | 6 | 6
ng/ml | 683 (147) | 521 (293) | 1239 (422)

ADVERSE EVENTS:
Time Frame: 30 days after end of treatment. Treatment ranged from 1 to 81 28-day cycles. The median number of cycles was 3.5 cycles.
Groups:
- Stratum A - 40 mg/Day: Patients on ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 40 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum A - 60 mg/Day: Patients on ritonavir-boosted or cobicistat-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum B - 60 mg/Day: Patients on efavirenz or etravirine-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum B - 100 mg/Day: Patients on efavirenz or etravirine-boosted antiretroviral therapy
  Patients receive cabozantinib s-malate 100 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
- Stratum C - 60 mg/Day: Patients who were on antiretroviral therapy that did not include the agents in stratums A or B, or were not on antiretroviral therapy.
  Patients receive cabozantinib s-malate 60 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
Arm/Group | Stratum A - 20 mg/Day | Stratum A - 40 mg/Day | Stratum A - 60 mg/Day | Stratum B - 60 mg/Day | Stratum B - 100 mg/Day | Stratum C - 60 mg/Day
All-Cause Mortality (participants affected / at risk) | 3/6 | 3/7 | 0/7 | 0/6 | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/7 | 5/7 | 3/6 | 1/3 | 2/7
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 7/7 | 6/6 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum A - 20 mg/Day (N=6) | Stratum A - 40 mg/Day (N=7) | Stratum A - 60 mg/Day (N=7) | Stratum B - 60 mg/Day (N=6) | Stratum B - 100 mg/Day (N=3) | Stratum C - 60 mg/Day (N=7)
atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
chest pain (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
pericardial tamonade (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
disease progression (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
fever (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
bronchial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Necrotizing fasciitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
skin infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0
small intestine infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 0 | 0 | 0
tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
arterial thromboembolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
MRSA (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum A - 20 mg/Day (N=6) | Stratum A - 40 mg/Day (N=7) | Stratum A - 60 mg/Day (N=7) | Stratum B - 60 mg/Day (N=6) | Stratum B - 100 mg/Day (N=3) | Stratum C - 60 mg/Day (N=7)
anemia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 1 | 1 | 1
TSH increased (Endocrine disorders) | 1 | 0 | 0 | 1 | 0 | 0
hypothyroidism (Endocrine disorders) | 2 | 2 | 3 | 1 | 0 | 2
blurred vision (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 0
constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 0 | 1
diarrhea (Gastrointestinal disorders) | 0 | 4 | 5 | 3 | 2 | 6
dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2
dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
gastroesophageal reflux (Gastrointestinal disorders) | 0 | 4 | 1 | 2 | 0 | 1
Gums bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
oral mucositis (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 1 | 1
nausea (Gastrointestinal disorders) | 2 | 4 | 5 | 4 | 0 | 5
oral pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1
proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
rectal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 2 | 0 | 3
chills (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
limb edema (General disorders) | 0 | 1 | 0 | 1 | 0 | 1
fatigue (General disorders) | 1 | 4 | 2 | 5 | 0 | 4
fever (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
flu like symptoms (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
night sweats (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
non cardiac chest pain (General disorders) | 0 | 0 | 2 | 1 | 0 | 0
pain (General disorders) | 2 | 1 | 1 | 1 | 0 | 1
gum infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0
Increased RPR titer (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
skin infection (Infections and infestations) | 0 | 1 | 2 | 2 | 0 | 0
upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
alanine aminotransferase increased (Investigations) | 3 | 3 | 3 | 2 | 1 | 3
increased alkaline phosphatase (Investigations) | 3 | 1 | 1 | 1 | 1 | 0
blood bilirubin increased (Investigations) | 2 | 0 | 2 | 0 | 0 | 0
LDH elevated (Investigations) | 1 | 2 | 0 | 0 | 1 | 0
increased creatinine (Investigations) | 2 | 0 | 1 | 1 | 0 | 1
INR increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
lipase increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0
lymphocyte count increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0
neutrophil count decreased (Investigations) | 3 | 2 | 2 | 1 | 2 | 4
lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0
platelet count decreased (Investigations) | 2 | 0 | 1 | 1 | 2 | 3
weight loss (Investigations) | 0 | 1 | 1 | 1 | 0 | 1
white blood cell decreased (Investigations) | 2 | 3 | 2 | 1 | 2 | 2
anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1 | 2
hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 1 | 1
hyperkalemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 0 | 0
hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 1 | 0
hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 2 | 0
hypocalcemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 1 | 2 | 1
hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 1 | 0
hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 1 | 1
hyponatremia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 4 | 0 | 1
hypophosphatemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 1 | 2 | 2
Elevated serum protein (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 1
bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
right knee strain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
myositis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
dizziness (Nervous system disorders) | 0 | 1 | 2 | 2 | 0 | 1
dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 2
headache (Nervous system disorders) | 0 | 2 | 1 | 1 | 0 | 1
paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2
peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 3 | 1 | 0 | 0
insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 1
hematuria (Renal and urinary disorders) | 1 | 0 | 2 | 2 | 0 | 0
proteinuria (Renal and urinary disorders) | 2 | 2 | 2 | 5 | 3 | 1
Ketones in urine (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0 | 0
renal calculi (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2 | 0 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
post nasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Elevated carbon dioxide (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0
dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 3
palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 4 | 5 | 1 | 1 | 2
pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
maculo-papular rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1 | 0 | 0
Hair graying (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0
skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1
hot flashes (Vascular disorders) | 0 | 2 | 2 | 0 | 0 | 0
hypertension (Vascular disorders) | 3 | 4 | 4 | 1 | 3 | 2
decreased eosinophils (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 1 | 0
Increased monocytes (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 0 | 0
Decrease Monocytes (Blood and lymphatic system disorders) | 0 | 3 | 2 | 1 | 1 | 0
Decreased RBC (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 1 | 0
Splenic and Kidney infarcts (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Stomach tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Altered bowel movement pattern (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Canker sores (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oral dysesthesia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Loss of balance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Elevated Urogilinogen (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bladder infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Shingles (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Periodontal disease (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Papulopustular Rash (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
aspartate aminotransferase increased (Investigations) | 3 | 4 | 3 | 3 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hemoglobin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
MCV elevated (Investigations) | 1 | 2 | 1 | 0 | 1 | 0
Elevated urea nitrogen (Investigations) | 1 | 0 | 1 | 1 | 0 | 0
Abnormal EKG (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Elevated PSA (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Elevated Neutrophils (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Elevated basophils (Investigations) | 1 | 1 | 1 | 1 | 0 | 0
Elevated serum protein (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 0 | 0
Elevated chloride (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 0
Decreased chloride (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Leukocyturia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0
Serum amylase increased (Investigations) | 0 | 1 | 1 | 2 | 1 | 0
Thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Left hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle cramp in legs (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Right peripheral vision loss (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Leucocyte in urine (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Bacteria in urine (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gynecological pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Increased urea nitrogen (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Decreased carbon dioxide (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nail coloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Increased sensitivity to heat and cold (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Poison ivy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Porokeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hair color lightening (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thromboemolic event (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Feels hot and cold (alternating) (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT01822522/Prot_SAP_000.pdf